CLINICAL TRIAL: NCT05451602
Title: Phase 1/2 Study of the Highly-selective RET Inhibitor,HEC169096 in Participants With Thyroid Cancer, Non-Small Cell Lung Cancer, and Other Advanced Solid Tumors
Brief Title: HEC169096 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEC169096-ST-101
Record Dates: First submitted 2022-07-03; First posted 2022-07-11 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-07

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HEC169096 (Experimental): Multiple doses of HEC169096
  Interventions: Drug: HEC169096

INTERVENTIONS:
Drug: HEC169096 — Multiple doses of HEC169096 during Phase 2；Oral dose of HEC169096 as determined during Phase 2.

SUMMARY:
An Open, Multi-Center Phase I/II Clinical Study To Evaluate The Safety, Tolerability, Pharmacokinetic Characteristics And Effectiveness Of HEC169096 In Patients With Thyroid Cancer, Non-Small Cell Lung Cancer, and Other Advanced Solid Tumors.

DETAILED DESCRIPTION:
This is an open-label, multi-center Phase 1/2 study in participants with advanced solid tumors, including RET fusion-positive NSCLC, MTC, and other tumors with RET activation. Phase I of this study includes a dose-escalation phase and a dose-expansion phase , which will focus on exploring MTD and/or RP2D of HEC169096 in patients with advanced solid tumours; Phase II will assess the efficacy and safety of HEC169096 at the RP2D dose.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1：Pathologically documented, definitively diagnosed non-resectable advanced solid tumor.
* Phase 2： All participants must have an oncogenic RET-rearrangement/fusion or mutation (excluding synonymous, frameshift, and nonsense mutations) solid tumor.
* Participants has Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2.
* Measurable or non-measurable disease as determined by RECIST 1.1;
* Adequate hematologic, hepatic and renal function;
* Life expectancy of at least 12 weeks;
* Negative pregnancy test (urine or serum) for female patients of childbearing potential;
* Participants agrees to provide tumor tissue (archived, if available or a fresh biopsy).

Exclusion Criteria:

* Participant's cancer has a known primary driver alteration other than RET.
* Nitrosourea, anthracyclines and mitomycin chemotherapy within 6 weeks prior to study treatment;
* Chemotherapy, immunotherapy, radiotherapy, or major surgery within 4 weeks or 5 half-lives (whichever is longer) prior to study treatment;
* Those who have received more than 30% of bone marrow radiation or wide-range radiotherapy within 4 weeks before the first study drug treatment (the patients receiving palliative radiotherapy are within 2 weeks before receiving study drug treatment);
* Had received traditional Chinese medicine for anti-tumor within a week before receiving study drug treatment;
* Had received live vaccine within 4 weeks prior to study treatment;
* Had received any investigational agent from other clinical study within 4 weeks or 5 half-lives (whichever is longer) prior to study treatment or are currently participating in other clinical trials;
* Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study treatment .
* Central nervous system (CNS) metastases or a primary CNS tumor that is associated with progressive neurological symptoms.
* Patients with other malignant tumors within 5 years before the first use of drugs
* Patients have a history of severe cardiovascular disease;
* Active hepatitis (Hepatitis B: HBsAg-positive and HBV-DNA ≥ 2000 IU/ mL or ≥ 10^4 cps/ mL; Hepatitis B: HCV antibody-positive and HCV-RNA positive), HIV antibody-positive.
* Patients with clinically active interstitial lung disease, active pneumonia, and radiation pneumonia requiring treatment;
* Poorly controlled pleural effusion, abdominal effusion, or pericardial effusion after intervention (such as drainage);
* Clinically significant active malabsorption syndrome or other diseases that may affect study drug administration and gastrointestinal absorption;
* Patients have been treated with any strong CYP3A inhibitors or inducers within 2 weeks prior to the first dose or PPIs in the first week before the first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: MTD and RP2D of HEC169096 | Cycle 1 (28 days) of treatment for MTD and at the end of every 2 cycle for RP2D for approximately 12 months or earlier if participant terminates from the study
  Determination of Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of HEC169096
Phase 2: Overall Response Rate | through study completion, an average of 1 year
  As assessed by Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)

CONTACTS AND LOCATIONS:
Locations (1):
- GuangDong Province Peoples Hospital, Guangzhou, China